CLINICAL TRIAL: NCT03200184
Title: Sofosbuvir and Daclatasvir in Treating Hepatitis C, A Study on 1000 Patients
Acronym: SD1000
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR.TUMS.DDRI.REC.1396.30
Record Dates: First submitted 2017-05-28; First posted 2017-06-27 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2017-05

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; sofosbuvir; daclatasvir
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Subjects will receive sofosbuvir and daclatasvir
  Interventions: Drug: sofosbuvir and daclatasvir

INTERVENTIONS:
Drug: sofosbuvir and daclatasvir — A fixed dose combination pill containing 400mg sofosbuvir and 60 mg daclatasvir given daily for 12 weeks. If a patient is cirrhotic, treatment duration would be 24 weeks.
  Other Names: Sovodak

SUMMARY:
The fixed-dose combination of sofosbuvir and daclatasvir in a single pill is being used for the treatment of hepatitis C in Iran. In this study the efficacy of this combination is evaluated in 1000 patient with hepatitis C.

DETAILED DESCRIPTION:
All cases of hepatitis C whether cirrhotic, post organ transplant, co-infected with HIV or hepatitis B, active drug abuse, on immune suppression and from all genotypes will be included. Patients will be treated by a single daily dose of a fixed-dose combination pill of 400mg sofosbuvir and 60 mg daclatasvir for 12 weeks. If a patient is cirrhotic, defined by liver stiffness > 12 kilopascal, either weight based ribavirin will be added or the treatment duration will be prolonged to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Positive qualitative hepatitis C virus RNA test on two occasions at least 6 months apart

Exclusion Criteria:

* Heart rate < 50/min,
* Taking amiodarone

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1448 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
The sustained viral response rate | 12 weeks after end of treatment
  Qualitative hepatitis C virus RNA polymerase chain reaction

SECONDARY OUTCOMES:
Adverse drug events | weeks 2, 4, 8, 12 and 24
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Reza Malekzadeh, MD, Study Chair — Tehran University of Medical Sciences
Locations (1):
- Shariati Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merat S; SD1000 Research Team. SD1000: High Sustained Viral Response Rate in 1361 Patients With Hepatitis C Genotypes 1, 2, 3, and 4 Using a Low-cost, Fixed-dose Combination Tablet of Generic Sofosbuvir and Daclatasvir: A Multicenter, Phase III Clinical Trial. Clin Infect Dis. 2020 May 6;70(10):2206-2212. doi: 10.1093/cid/ciz628. PMID 31504303